CLINICAL TRIAL: NCT01647698
Title: Beyond the Physical: Enhancing Psychosocial Functioning in Parkinson's Disease
Brief Title: Pilot Study to Determine if Working Memory Training Aids Cognitive Functioning in Patients With Parkinson's Disease
Acronym: PDWM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gail Eskes (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Gail Eskes, Dr. Gail Eskes, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PDWM-2012-07
Record Dates: First submitted 2012-07-13; First posted 2012-07-23 (Estimated); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; near transfer; far transfer; working memory; fluid intelligence; cognitive training; dual n-back
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Early training group (Experimental): The early training group will consist of 10 randomly assigned participants who will begin the adaptive working memory training task immediately after baseline assessment. They will continue training on the adaptive working memory training task for 5 weeks, after which they will continue for 5 weeks using a non-adaptive working memory task (active control task).
  Interventions: Behavioral: Adaptive working memory training task; Behavioral: Non-adaptive working memory training task (i.e. an active control task)
- Late training group (Experimental): The late training group will consist of 10 randomly assigned participants who will engage in a non-adaptive working memory training task (i.e. an active control task) immediately after baseline assessment for 5 weeks. After the initial 5 weeks of the active control task they will then switch to the adaptive working memory task (the intervention) for 5 weeks. This is a randomized controlled cross-over design.
  Interventions: Behavioral: Adaptive working memory training task; Behavioral: Non-adaptive working memory training task (i.e. an active control task)
- No training group (Placebo Comparator): The no training group will engage in no training over the course of the pilot study, but will still participate in baseline, 5 week, 10 . This will allow us to determine if changes in the outcome and assessment variables are due to the working memory training or progression in the disease itself.
  Interventions: Behavioral: No training

INTERVENTIONS:
Behavioral: Adaptive working memory training task — The working memory training task will consist of an adaptive working memory computer program that will test and extend patients' working memory capacity.
  Adaptive refers to the increase in the number of items that the patient is required to remember.
  Arms: Early training group; Late training group
Behavioral: Non-adaptive working memory training task (i.e. an active control task) — Active control task will consist of a non-adaptive working memory task.
  Arms: Early training group; Late training group
Behavioral: No training — No training during the experiment.
  Arms: No training group

SUMMARY:
This project will investigate the feasibility and preliminary effectiveness of an intensive and focused working memory training program for patients in the early stages of PD receiving dopaminergic therapy. The investigators hypothesize that working memory training will be an effective method of improving working memory and related cognitive and behavioural functions in PD patients.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is not an exclusively motor disease; more than half of individuals with PD experience cognitive impairment even in the early stages of the disease and many develop dementia as the disease progresses. As a result, attention, memory, planning and organizational skills can be affected, interfering with everyday functioning (e.g. shopping, managing finances, job skills). Thus, interventions to improve cognitive abilities are needed to enhance psychosocial function and overall quality of life.

Some cognitive deficits, such as problems with working memory, are apparent even in the early stages of the disease. Working memory (WM) is the ability to actively maintain and manipulate information in one's mind and is needed for many complex tasks such as learning, communication and problem-solving . Individuals with PD often show deficits in both WM maintenance (e.g., holding a phone number in mind to make a call) and manipulation (e.g.,mental calculation at the grocery store checkout) skills, depending upon the stage of the disease and progression of damage to frontal-subcortical circuits. Attempts to identify pharmacological agents that ameliorate cognitive dysfunction have been largely unsuccessful or associated with undesirable side effects (e.g. Vale, 2009).

The investigators propose that specific cognitive training to improve WM could provide direct benefit to psychosocial function of PD patients; it could potentially enhance any positive benefits or reduce the negative effects of pharmacological treatment without an added risk of side effects as well. Promising interventions focused on intensive and direct WM training are emerging and have been shown to generalize to other cognitive domains, such as fluid intelligence.

Cognitive training has been successful in patients with traumatic brain injury, who also show WM deficits as a result of damage to frontal-subcortical circuits. In addition, successful WM training is associated with changes in dopamine receptor density as well as changes in patterns of neural activity in task-relevant areas of the brain. To date, a limited number of small group studies provide preliminary evidence that some aspects of cognitive function can be enhanced by training in PD patients also receiving dopaminergic therapy, although few use control groups to account for potential repeated testing practice effects.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of idiopathic Parkinson's disease
* self-reported concerns about their working memory, or working memory deficits that were identified by a clinical examination
* be classified as Hohn & Yahr Stage 1 or 2
* be receiving a stable dose of dopaminergic therapy

Exclusion Criteria:

* presence of dementia or other significant neurological or psychiatric conditions, as determined by clinical history
* Classification as Hohm & Yahr Stage 3 or 4
* Not on a stable dos of dopaminergic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline Working memory function | baseline
  Working memory will be measured using the operation span task, the symmetry span task and the Sternberg memory scanning tasks.
  Operation span - This is a dual-task in which participants complete mathematical reasoning (e.g. solving a mathematical equation) while using short-term verbal memory to remember words.
  Symmetry span: This is a dual task in which participants discriminate about the symmetry of visual stimuli while using short-term spatial memory to remember the locations of stimuli.
  Sternberg memory scanning task - number memory test
Change in working memory function between baseline and 5 weeks post training onset | 5 weeks post training onset
Change in working memory function between baseline and 10 weeks post training onset | 10 weeks post training onset
Change in working memory function between baseline and 22 weeks post training onset | 22 weeks post training onset

SECONDARY OUTCOMES:
Baseline fluid intelligence | Baseline
  Fluid intelligence will be measured using Cattell's Culture Fair Intelligence Test, a measure of analogical reasoning, and Raven's Progressive Matrices, a measure of spatial reasoning.
change in fluid intelligence between baseline and 5 weeks post training onset | 5 weeks post training onset
Change in fluid intelligence between baseline and 10 weeks post training onset | 10 weeks post training onset
Change in fluid intelligence between baseline and 22 weeks post training onset | 22 weeks post training onset
Baseline Executive functioning | Baseline
  Executive functioning will be measured using the Dysexecutive Questionnaire. It is a self-report and other-report of everyday behaviours reflecting executive function.
Change in executive functioning between baseline and 5 weeks post training onset | 5 weeks post training onset
Change in executive functioning between baseline and 10 weeks post training onset | 10 weeks post training onset
Change in executive function between baseline and 22 weeks post training onset | 22 weeks post training onset

CONTACTS AND LOCATIONS:
Overall Officials: Gail Eskes, PhD, Study Director — Dalhousie University; Raymond Klein, PhD, Study Chair — Dalhousie University; David Westwood, PhD, Study Chair — Dalhousie University; Stephanie Jones, PhD, Principal Investigator — Dalhousie University
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada